CLINICAL TRIAL: NCT02427880
Title: Acetazolamide and Hydrochlorothiazide Followed by Furosemide Versus Hydrochlorothiazide and Furosemide Followed by Furosemide for the Treatment of Adults With Refractory Nephrotic Edema: A Randomized, Double-Blind Trial
Brief Title: Role of Acetazolamide and Hydrochlorothiazide Followed by Furosemide in Treating Nephrotic Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Amin Fallahzadeh, MD-MPH, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7308
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Nephrotic Syndrome; Edema
Keywords: Edema; Nephrotic syndrome; Acetazolamide; Furosemide
MeSH Terms: conditions — Nephrotic Syndrome; Edema | interventions — Acetazolamide; Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental): Each patient receives 250 mg of acetazolamide and 50 mg of hydrochlorothiazide daily for 1 week. Then they are prescribed 40 mg of furosemide daily for 2 weeks.
  Interventions: Drug: Acetazolamide and Hydrochlorothiazide Followed by Furosemide
- Furosemide (Active Comparator): Each patient is prescribed 40 mg of furosemide and 50 mg of hydrochlorothiazide daily for 1 week. Then they receive 40 mg of furosemide daily for 2 weeks.
  Interventions: Drug: Furosemide and Hydrochlorothiazide Followed by Furosemide

INTERVENTIONS:
Drug: Acetazolamide and Hydrochlorothiazide Followed by Furosemide
  Other Names: Diamox Sequels and Microzide Followed by Lasix
  Arms: Acetazolamide
Drug: Furosemide and Hydrochlorothiazide Followed by Furosemide
  Other Names: Lasix and Microzide Followed by Lasix
  Arms: Furosemide

SUMMARY:
The purpose of this study is to determine whether using furosemide following acetazolamide is effective in treating refractory edema associated with nephrotic syndrome.

DETAILED DESCRIPTION:
Edema is referred to increase in interstitial fluid that is clinically evident. The main causes of generalized edema are heart failure, renal failure, nephrotic syndrome, glomerulonephritis and chronic liver failure. In some cases, edema is treated by management of the underlying disease. However, in some other cases edema may persist and become more severe that needs adjuvant treatments. Because use of diuretics such as furosemide and hydrochlorothiazide is not completely effective in treating severe refractory edema, use of some other diuretics is also recommended. In this double-blind clinical trial, weight and some lab data including blood urea nitrogen, serum creatinine, serum sodium, serum potassium, serum albumin, urine sodium, urine potassium, 24-hour urine volume, 24-hour urine protein and 24-hour urine creatinine of 20 random adult patients with nephrotic syndrome who have refractory edema and GFR>60 ml/min/1.73m2 and are referred to nephrology clinic of Shiraz University of Medical Sciences will be measured; the patients should not have hypokalemia and other causes of edema such as heart failure or cirrhosis. Then the patients are divided into 2 groups with 10 members in each. The first group will be prescribed 40 mg of furosemide and 50 mg of hydrochlorothiazide and the second one will receive 250 mg of acetazolamide and 50 mg of hydrochlorothiazide daily for 1 week. Then, weight and mentioned lab data will be measured again. After that, all the patients will have 40 mg of furosemide daily for 2 weeks. Then, weight and mentioned lab data will be measured for one more time.

ELIGIBILITY:
Inclusion Criteria:

1. Having refractory edema due to nephrotic syndrome
2. Having GFR>60 ml/min/1.73m2
3. Being able to come for weekly visit
4. Having the minimum age of 18 years
5. Signing the informed consent form

Exclusion Criteria:

1. Hypokalemia
2. Pregnancy
3. Renal transplant
4. active malignancy or infection
5. acidosis
6. Using NSAIDs
7. Having another causes of edema including liver cirrhosis, heart failure
8. Neurologic or psychiatric problem hindering adherence to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight at the end of third week | Baseline and at the end of the third week

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure at the end of third week | Baseline and at the end of the third week
Change from baseline in serum sodium at the end of third week | Baseline and at the end of the third week
Change from baseline in serum potassium at the end of third week | Baseline and at the end of the third week
Change from baseline in blood urea nitrogen at the end of third week | Baseline and at the end of the third week
Change from baseline in serum creatinine at the end of third week | At the start and at the end of the third week
Change from baseline in serum albumin at the end of third week | Baseline and at the end of the third week
Change from baseline in urine sodium at the end of third week | Baseline and at the end of the third week
Change from baseline in urine potassium at the end of third week | Baseline and at the end of the third week
Change from baseline in 24-hour urine volume at the end of third week | Baseline and at the end of the third week
Change from baseline in 24-hour urine creatinine at the end of third week | Baseline and at the end of the third week
Change from baseline in 24-hour urine protein at the end of third week | Baseline and at the end of the third week

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mahdi Sagheb, MD, Study Chair — Nephrologist at Shiraz University of Medical Science

REFERENCES:
- [Background] Soleimani M. A novel target for diuretic therapy. Iran J Kidney Dis. 2012 Nov;6(6):419-25. PMID 23146978